CLINICAL TRIAL: NCT02509572
Title: Improvement of STI Detection in Adolescent Emergency Department Patients
Acronym: SHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Monika Goyal, Assistant Professor of Pediatrics & Emergency Medicine, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00004169
Record Dates: First submitted 2015-07-21; First posted 2015-07-28 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Sexually Transmitted Infections
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Support Arm (Experimental): Patients randomized to the intervention will complete a sexual health screen (SHS). The results of the SHS will provide decision support for STI testing by risk stratifying patients with screening recommendations to the clinician based on risk.
  Interventions: Behavioral: Sexual health screen (SHS)
- Usual Care Arm (No Intervention): Patients randomized to the usual care arm will complete the sexual health screen (SHS). However these results and the STI testing decision support will not be shared with the clinician.

INTERVENTIONS:
Behavioral: Sexual health screen (SHS) — Decision support for STI screening through a novel sexual health screen
  Arms: Decision Support Arm

SUMMARY:
The goal of this trial is to test a novel means of collecting patient-entered sexual health information for the provision of clinical decision support to increase the testing and detection of sexually transmitted infections (STI) in adolescent emergency department (ED) patients at high risk for STIs.

DETAILED DESCRIPTION:
The investigators have developed a novel means of collecting sexual health information from adolescents in the emergency department (ED) through the use of an audio-computer assisted self-interview (ACASI). This information can then be used to provide clinical decision support to clinicians for targeted sexually transmitted infection (STI) screening in the ED for adolescents. This randomized trial randomizes patients to whether or not the clinician receives the decision support and tests whether provision of decision support results in increased STI screening for patients who report high risk sexual activity. Secondary outcomes include evaluation of whether the clinical decision support results in increased STI detection, and identifying factors associated with adapting the clinical decision support.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-19 presenting to the emergency department.

Exclusion Criteria:

* history of developmental delay,
* medical instability,
* altered mental status,
* unable to understand English

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 720 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with difference in frequency of STI testing between the ACASI-SHS group compared to the usual care group. | an expected average of 4-6 hours.

SECONDARY OUTCOMES:
The proportion of adolescents who test positive for an STI in the intervention group in comparison to the usual care group. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Monika Goyal, MD, MSCE, Principal Investigator — CNMC
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Goyal MK, Fein JA, Badolato GM, Shea JA, Trent ME, Teach SJ, Zaoutis TE, Chamberlain JM. A Computerized Sexual Health Survey Improves Testing for Sexually Transmitted Infection in a Pediatric Emergency Department. J Pediatr. 2017 Apr;183:147-152.e1. doi: 10.1016/j.jpeds.2016.12.045. Epub 2017 Jan 10. PMID 28081888